CLINICAL TRIAL: NCT01553773
Title: Hyaluronic Acid Concentration in Postmenopausal Facial Skin After Estradiol and Genistein Topical Treatment: Double-blind and Randomized Clinical Trial of Efficacy
Brief Title: Postmenopausal Facial Skin After Estradiol and Genistein Topical Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Marisa T Patriarca, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIFESPMP#1
Record Dates: First submitted 2012-03-05; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Atrophy
Keywords: Hyaluroic acid; Estradiol; Isoflavone; Skin; Postmenopause
MeSH Terms: conditions — Atrophy | interventions — Isoflavones; Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoflavone (Experimental): a gel with isoflavones (genistein 4%)
  Interventions: Drug: isoflavone
- Estradiol (Experimental): gel with 17-β estradiol 0.01%
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: isoflavone — treatments: a gel with 17-β estradiol 0.01% (n = 15) and a gel with isoflavones (genistein 4%). The gels were applied once per day. the lenght of treatment was 24 weeks.
  Other Names: Group G
  Arms: Isoflavone
Drug: Estradiol — a gel with 17-β estradiol 0.01%. Once per day. The lenght of treatment was 24 weeks.
  Other Names: Group E
  Arms: Estradiol

SUMMARY:
The aim of this trial was to compare the effects of estradiol or genistein treatment on the hialuronic acid concentration on the postmenopausal facial skin. In this study, 30 postmenopausal women were evaluated through a prospective, randomized, double-blind trial. The volunteers were postmenopausal women treated in the Gynecology Department of the Federal University of São Paulo (UNIFESP). The participants were divided into two groups: group E, treated with 17 β estradiol gel 0.01% (n = 15), and group G, treated with genistein gel 4 % (isoflavones, n=15). The length of treatment was 24 consecutive weeks. Preauricular skin biopsies were performed on each patient before and after the treatment for evaluating hyaluronic acid in the tissue. The materials were processed through immunohistochemical and biochemical methods.

DETAILED DESCRIPTION:
Postmenopausal volunteers were recruited in Brazil from the Endocrinological Gynecology Division of the Gynecology Department of Federal University of São Paulo (UNIFESP). All women participated in this prospective, randomized, double-blind and estrogen-controlled study and approved by the local Ethics and Research Committee (Report No 386/2004). The evaluation of all of the subjects consisted of a detailed history, a physical exam, and a laboratory workup. The study protocol was approved by the UNIFESP School of Medicine Human Investigation Committee, and every participant had to provide written informed consent before enrollment.

Intervention Independent pharmacists dispensed either isoflavone or estrogen containers according to a computer-generated randomization list. The containers, as well as a jar for treatments, had identical appearance and color. The researchers were responsible for seeing the women allocated the next available number on entry into the trial, and each woman collected her containers directly from the pharmacy department. The code was revealed to the researchers once recruitment, data collection, and histological analyses were complete. If a health problem occurred, an independent physician who was blinded to the patient's treatment group examined her. If necessary, this physician prescribed laboratory exams for exclusion of any serious systemic side-effects. A number two punch biopsy of facial skin from the preauricular area was performed before and after the 24-week gel treatment. The women applied the gel on their facial skin daily at night, and in the morning, they used a gel sunscreen only. They were advised not to use any other cream. To assess possible systemic hormonal effects, hormonal vaginal cytology samples were taken at all visits (baseline and after 6, 12, 18, and 24 weeks of treatment) and estradiol blood samples before and after the treatment.

Groups The participants flowed through each stage of the study. After the end of study, the label was opened, and the treatment groups with the same number were classified. Fifteen patients were required for each study group: group E, treated with a gel with 17-β estradiol 0.01% (n = 15), and group G, treated with a gel with isoflavones (genistein 4%) (n = 15).

Processing of the material After the collection, the biopsies were immediately fixed for 24 hours in 10% formaldehyde solution and then processed for paraffin via dehydration in ethanol in increasing concentrations, diaphanization in xylol and impregnation by liquid paraffin in drying oven set at a temperature of 60 °C (methodology recommended by Michalany, 1998). The paraffin blocks were submitted to cuts of 3 μm with a Minot microtome. The cuts for immunohistochemistry were placed on slides previously treated with silane to 5 % and brought to oven at 37 °C for 24 hours for drying. Additionally, sections were made of 20 μm and placed in tubes of 2ml for the biochemical processing.

ELIGIBILITY:
Inclusion Criteria:

* two to five years postmenopause;
* FSH > 40 mU/ml;
* estrogen levels < 20 pg/ml;
* body mass index (BMI) < 30 kg/m2

Exclusion Criteria:

* treatment with estrogens or soybeans for the previous 12 months;
* tobacco user;
* women who had a contraindication for hormone therapy, who had been using retinoids or herbal substances, and those who had a history of collagen diseases.
* also, strict vegetarianism, high fiber- or high soy-diet consumption;
* regular consumption of vitamin and mineral supplementation greater than the Recommended Dietary Allowances;
* antibiotic treatment;
* a history of chronic disorders, including endocrine or gynecological diseases or neoplasia, as well as benign breast disease; and
* regular use of medication known to interfere with the study endpoints.
* patients with cervico-vaginal cytology classified as Papanicolaou Class III or more were also excluded.
* participants with hypertension who were using two or more antihypertensive drugs were not included in this study.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Analysis of hyaluronic acid concentration in postmenopausal facial skin | up to 6 months
  A number two small punch biopsy of facial skin from the preauricular area was performed before and after the 24-week gel treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa T Patriarca, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Department of Gynecology - UNIFESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva LA, Ferraz Carbonel AA, de Moraes ARB, Simoes RS, Sasso GRDS, Goes L, Nunes W, Simoes MJ, Patriarca MT. Collagen concentration on the facial skin of postmenopausal women after topical treatment with estradiol and genistein: a randomized double-blind controlled trial. Gynecol Endocrinol. 2017 Nov;33(11):845-848. doi: 10.1080/09513590.2017.1320708. Epub 2017 May 16. PMID 28508697